CLINICAL TRIAL: NCT04371341
Title: A Comparative Study Between Different Local Anesthetic Volumes Injected During Erector Spinae Block to Reduce Postoperative Opioid Consumption in Patients Undergoing Open Simple Nephrectomy Operations; a Randomized Controlled Trial
Brief Title: A Comparative Study Between Different Volumes During Erector Spinae Block for Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: _MD-248-2019
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Pain Management
Keywords: erector spinae; -block; volume; pain
MeSH Terms: conditions — Bites and Stings; Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: 4 groups with 20 patients for each group where group C will not receive erector spinae block and so will be the control group while groups which will receive erector spinae block will be E1,E2,E3 and will receive 0.25% bupivacaine with volumes of 2.5,3.4,6.6 ml/segment respectively.
Who Masked: Care Provider, Investigator
Masking Description: the care provider and investigator will be masked from the volume injected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- E1 (Experimental): will receive erector spinae block with 0.25% bupivacaine volume of 2.5 ml/segment
  Interventions: Procedure: erector spinae block by 0.25% bupivacaine
- E2 (Experimental): will receive erector spinae block 0.25% bupivacaine with volume of 3.4ml/segment
  Interventions: Procedure: erector spinae block by 0.25% bupivacaine
- E3 (Experimental): will erector spinae block receive 0.25% bupivacaine with volume of 6.6 ml/segment
  Interventions: Procedure: erector spinae block by 0.25% bupivacaine
- C (No Intervention): will not receive erector spinae block

INTERVENTIONS:
Procedure: erector spinae block by 0.25% bupivacaine — A mark will be applied on the required level (T8), the midline (spinous processes) and the injection points 3 cm from midline.While the patient is in a sitting position with support from a member of staff, Preparation of the field with iodine will be made. Using ultrasound guidance with a 6-10 MHz linear probe anatomical landmarks will be identified including the transverse process at T8 level and the three layers of muscles from posterior to anterior: trapezius-rhomboid-erector spinae. After subcutaneous lidocaine 2% injection a 22-G spinal needle will be inserted under ultrasound guidance in plane, aiming towards the transverse process. After a Gentle contact with the transverse process, 0.25% bupivacaine is injected in increments with careful repetitive aspiration to avoid intravascular injection.
  Other Names: erector spinae plane block
  Arms: E1; E2; E3

SUMMARY:
Since its first description by Forero et al. there have been many articles and case reports including an increasingly number of indications for the ESP block: chronic and acute pain treatment, rib fractures management in the emergency setting, treatment of abdominal surgical pain, hip arthroplasty , analgesic management in breast surgery,or in spinal surgery.Although ESP block successfully reduced postoperative opioid consumption in clinical reports, no studies thus have investigated the optimum volume of bupivacaine for ESP block as regard a review of the medical literature on December 27th, 2017 that searched terms in 14 articles clearly stated the volume of the bolus and the spread of the anesthetic after an injection of LA, the volume needed to cover one dermatome widely varies from 2.5 mL to 6.6 mL, with a median value of 3.4 mL. Furthermore, the maximum number of dermatomes reached by a single bolus in ESP was of 9 dermatomes after a 30 mL bolus.

Thus, in this study, the investigators evaluate the effect of ESP block which will be performed by using three different volumes (2.5, 3.4 ,6.6 ml/segment) of bupivacaine with the same concentration ,technique ,site of injection and operation.

DETAILED DESCRIPTION:
INTRODUCTION In recent years a number of important fascial plane blocks have been described blocking the dorsal, lateral and anterior cutaneous nerves of the thorax and abdome].The advantage common to all of these blocks is that they are technically easier to perform with lower risk for serious complications.Since its first description by Forero et al. there have been many articles and case reports including an increasingly number of indications for the ESP block: chronic and acute pain treatment , rib fractures management in the emergency setting , treatment of abdominal surgical pain , hip arthroplasty , analgesic management in breast surgery ,or in spinal surgery.The ESP block targets the erector spinae plane, which lies in the chest wall between the anterior surface of the cephalo caudal oriented erector spinae muscles and the posterior surface of the spinal transverse processes. LA is deposited in the fascial plane deep to the erector spinae muscle and superficial to the tips of the transverse processes, from where it diffuses to the dorsal and ventral rami of spinal nerves, achieving an extensive multi-dermatomal sensory block of the posterior, lateral, and anterior thoracic wall .Chin et al reported that an injection of 20 ml into the ESP produces clinical and radiographic evidence of spread that extends at least three vertebral levels cranially and four levels caudally from the site of injection.A study with magnetic resonance imaging demonstrated and confirmed that its mechanism of action is likely linked to the transforaminal and epidural spread, which may be a potential advantage because the ESP block provides abdominal visceral analgesia unlike the others .beside its ability to spread to paravertebral and intervertebral spaces and ability to block the sympathetic nerve fibers. the ESP block is considered as a peri-paravertebral regional anesthesia technique.LAs, is injectted with volumes ranging from 20 mL to 40 mL, and concentrations ranging from 0.25%-0.5%.even though a higher LA concentration might allow for better diffusion into the paravertebral space .

Open surgery remains common for patients requiring radical or partial nephrectomy and is associated with a high incidence of intense immediate postoperative pain and chronic pain in the months following surgery. ESP block was for open partial nephrectomy with excellent results both in the intraoperative and postoperative period, with a large reduction in the use of opioids.

Although ESP block successfully reduced postoperative opioid consumption in clinical reports, no studies thus have investigated the optimum volume of bupivacaine for ESP block as regard a review of the medical literature on December 27th, 2017 that searched terms in 14 articles clearly stated the volume of the bolus and the spread of the anesthetic after an injection of LA, the volume needed to cover one dermatome widely varies from 2.5 mL to 6.6 mL, with a median value of 3.4 mL. Furthermore, the maximum number of dermatomes reached by a single bolus in ESP was of 9 dermatomes after a 30 mL bolus.

Thus, in this study, the investigators evaluate the effect of ESP block which will be performed by using three different volumes (2.5, 3.4 ,6.6 ml/segment) of bupivacaine with the same concentration ,technique ,site of injection and operation.

Methodology:

Eighty Patients, aging from 18-50 years with ASA physical status I and II, undergoing open simple nephrectomy will be included and randomly distributed into 4 groups with 20 patients for each group where group C will not receive erector spinae block and so will be the control group while groups which will receive erector spinae block will be E1,E2,E3 and will receive 0.25% bupivacaine with volumes of 2.5,3.4,6.6 ml/segment respectively.

The day before surgery, all patients will be instructed to fast for 6-8 hours. On the day of the operation,the patient will arrive to the preparation room 1 hour before operation,to allow time for the block procedure and a minimum of 45 minutes after the block to pass, an 18 G cannula insertion, a start of IV fluid drip, and premedication with 0.02-0.03 mg/kg intravenous midazolam will be done. All basic monitoring will be applied (ECG/HR/SpO2/NIBP), and baseline values for HR, SPO2 ,SBP,DBP and MAP will be documented then every 5 minutes till the patient reaches the operating room.

A mark will be applied on the required level (T8), the midline (spinous processes) and the injection points 3 cm from midline.While the patient is in a sitting position with support from a member of staff, Preparation of the field with iodine will be made. Using ultrasound guidance with a 6-10 MHz linear probe anatomical landmarks will be identified including the transverse process at T8 level and the three layers of muscles from posterior to anterior: trapezius-rhomboid-erector spinae. After subcutaneous lidocaine 2% injection a 22-G spinal needle will be inserted under ultrasound guidance in plane, aiming towards the transverse process. After a Gentle contact with the transverse process, the volume of 0.25% bupivacaine will be injected according to each group 2.5, 3.4 ,6.6 ml/segment in increments with careful repetitive aspiration to avoid intravascular injection.

Spread of the local anesthetic will be monitored by U/S anterior to erector spinae muscles (dividing erector spinae muscles from transverse process with caudal and cephalic spread) then the end point of local anesthetic will be marked and the corresponding covered level will be assessed caudal and cephalic from T8.onset of the block will be tested by pin brick test every 10 minutes after performing the block maximum 30 minutes otherwise it will be considered failed block and documented for each group while dermatomal spread will be assessed by pin brick test 30 minutes after onset of the block and will be documented.

Then the patient will be transferred to the OR. All basic monitoring will be applied (ECG/HR/SpO2/NIBP) while monitoring of end-tidal CO2, neuromuscular block and depth of anesthesia using Bispectral index (BIS) monitor will be initiated after induction of anesthesia and values will be recorded for HR, SPO2 ,SBP,DBP ,MAP and ETCO2 every 5 minutes till the end of the surgery then for 30 minutes from time of reaching PACU.

General anesthesia will be inducted with 2 mg/kg propofol, 1μg/kg fentanyl and 0.5 mg/kg atracurium to facilitate endotracheal intubation. After intubation the lungs will be mechanically ventilated to maintain the ETCO2 35-40 mmHg. Then Patient positioned in the lateral position. Anesthesia will be maintained with isoflurane keeping the ET concentration of isoflurane 1-2% to maintain the BIS value 40-60. Atracurium besylate top-up doses 0.1mg/kg will be given based on the response to train of four ulnar nerve stimulation. Additional fentanyl dose of 0.5 µg/kg IV for maximum of 2 µg/kg will be given if HR and or BP increased more than 20% from baseline in response to surgical stimulation and the total dose of fentanyl will be recorded.

The patient's pain will be monitored and documented using the Numerical Rating Score (NRS) for pain at times 0,30 minutes, 1, 2, 4, 6, 8, 10, 12, 18 and 24 hours. The "zero" point of time will be the moment the patient recovered from general anesthesia. Time to first analgesic requirement will be recorded. Rescue medication for pain will be given on demand including 1 g paracetamol IV when NRS >/= 2 but < 4 and if NRS is 4 or more a 5 mg morphine IV with maximum dose of 10 mg every 6 hours and the total consumption of these medications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-50 years with ASA I-II undergoing open simple nephrectomy operation.

Exclusion Criteria:

* Cardiovascular disease.
* Cerebrovascular insufficiency.
* Coagulation defects.
* hepatic insufficiency.
* Hypersensitivity to the study drugs.
* Pregnant patient. And patients receiving vasoactive drugs or beta blockers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption in milligrams in the three groups | 24 hours
  if NRS is 4 or more a 5 mg morphine IV with maximum dose of 10 mg every 6 hours will be given and the total consumption of these medications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Omar, M.D., Study Director — Cairo University
Locations (1):
- anesthesia department at Cairo University, Cairo, Elmanial, Egypt

IPD SHARING:
Plan to Share IPD: No
introduction and methodology are to be shared

REFERENCES:
- [Background] 1. Forero M, Adhikary SD, Lopez H, Tsui C,Chin KJ. The Erector Spinae Plane Block:A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med 2016 ;41(5):621-7. 2. Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth 2017;118(3):474-5 3. Josh Luftig P, Mantuani D, Herring AA, Dixon B, Clattenburg E, Nagdev A. The authors reply to the optimal dose and volume of local anesthetic for erector spinae plane blockade for posterior rib fractures. Am J Emerg Med 2018;36(6):1103-4 4. Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia 2017;7(4):452-60 5. Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth 2018;47:5-6